CLINICAL TRIAL: NCT03306849
Title: Ultrasonographic Evaluation of Anovulatory Disorders in Lean and Overweight Women
Status: Completed | Type: Observational
Sponsor: Cornell University (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 1410015577
Record Dates: First submitted 2017-10-06; First posted 2017-10-11 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Menstrual Cycle Abnormal; PCOS; Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — 26mL Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Regular menstrual cycles: Women will be assigned to this category if they report a history of regular menstrual cycles (every 21 to 35 days). Recruitment will be targeted such that equal numbers of lean (BMI <25kg/m2) and overweight or obese (BMI >24.9kg/m2) participate.
- Normoandrogenic anovulation: Women will be assigned to this category if they do not have clinical or biochemical androgen excess and report a history of irregular menstrual cycles (<21 days or >35 days), including women with a pre-existing diagnosis of PCOS. Recruitment will be targeted such that equal numbers of lean (BMI <25kg/m2) and overweight or obese (BMI >24.9kg/m2) participate.
- Hyperandrogenic anovulation: Women will be assigned to this category if they have clinical or biochemical androgen excess and report a history of irregular menstrual cycles (<21 days or >35 days), including women with a pre-existing diagnosis of PCOS. Recruitment will be targeted such that equal numbers of lean (BMI <25kg/m2) and overweight or obese (BMI >24.9kg/m2) participate.

SUMMARY:
The investigators would like to determine whether ultrasound features of the ovaries can be used to reliably diagnose different types of anovulatory disorders in women across all body types. The study will also try to establish whether ultrasound features of the ovary can reflect the degree of reproductive and metabolic problems that a woman with irregular or absent periods might be experiencing.

DETAILED DESCRIPTION:
This study is being conducted in order to determine if ultrasound features of the ovaries can be used to reliably diagnose different types of anovulatory disorders in women across all body types. The study will also try to establish whether ultrasound features of the ovary can reflect the degree of reproductive and metabolic problems that a woman with irregular or absent periods might be experiencing. In this way, the researchers can help to maximize the information that can be received when using ultrasound to evaluate patients with concerns over irregular menstrual cycles and/or infertility.

The ovaries are the site of egg production and normally release one egg every month. The process of releasing an egg is called ovulation. The act of releasing an egg is the body's way of ensuring a woman's fertility each month during her reproductive years. There are a number of reasons why ovulation may not occur regularly in women. Some of these reasons are believed to relate to male hormone production (i.e. androgens), body composition, nutrition and overall metabolic health. However, the precise ways in which these factors affect ovulation are unknown.

The researchers plan to evaluate how the ovaries look and function in a large group of women. Their goal is to recruit both lean and overweight women to this study and include both women that have regular, predictable menstrual cycles as well as those that have infrequent or absent menstrual cycles. The researchers will include women with irregular cycles due to increased androgen production, or hyperandrogenic anovulation - as well as those that have irregular cycles but normal androgen levels or normoandrogenic anovulation. The researchers will use ultrasound to collect information on how the ovaries look and function, and then relate the features of the ovaries to body composition, reproductive and metabolic hormones as well as nutritional factors. Because features of the ovaries are expected to be different in lean and overweight women, the researchers hope to develop ultrasound criteria that will help healthcare providers to diagnosis specific ovulation problems in women across all body sizes. Together, this research will help to better understand the complex relationship between nutrition, metabolism and reproductive health in women.

To accomplish these objectives, the investigators plan to recruit 50 women with regular menstrual cycles, 50 women with normoandrogenic anovulation, and 50 women with hyperandrogenic anovulation. Their goal is to recruit an equal number of women in each group who are lean (BMI; Normal weight = 18.5 - 24.9 kg/m2) and overweight or obese (BMI; Overweight = 25 - 29.9 kg/m2; Obese >= 30kg/m2). Ultrasound scans of the ovaries will be assessed for the total number, size, and distribution of follicles using both two- and three-dimensional imaging techniques. Participants will have blood samples collected determine serum concentrations of luteinizing hormone (LH), follicle stimulating hormone (FSH), estradiol, progesterone. The following metabolic parameters will be assessed: (1) 75-gram oral glucose tolerance test to characterize glucose and insulin dynamics at 0, 30, 60, 90, and 120 minutes post-glucose ingestion; (2) dual X-ray absorptiometry (DXA) scan to quantify body fat and lean muscle distribution; (3) vitals and anthropometry assessment to measure waist and hip circumference, height, weight, blood pressure, and heart rate, and (4) fasting blood tests to detect serum concentrations of androgens (i.e., total testosterone, androstenedione, free androgen index) and serum markers of metabolic syndrome (i.e., lipids and hemoglobin A1C). Participants will complete a food frequency questionnaire and physical activity questionnaire. A researcher may also provide participants with an accelerometer to wear for a week.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-45 years
* At least 2y post-menarche
* BMI >18.5kg/m2
* Good visibility of the ovaries on ultrasound

Either:

* Regular menstrual cycles (21-35 days);
* Irregular menstrual cycles (>35 days); or
* Previous diagnosis of PCOS from a primary care provider

Exclusion Criteria:

* Weight >300lbs
* Currently pregnant or breast feeding
* History of ovarian surgery
* Use of medications or supplements known or suspected to interfere with reproductive function and/or glucose and lipid metabolism in the past 3 months
* Evidence of reproductive aging as assessed by the principal criteria of STRAW+10 stages

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women must be able to transport to Weill Cornell University. Eligible participants are between 18-45 years with a BMI of 18.5 kg/m2 or higher. Women are screened and enrolled following consent based on their response to our advertisements. Women are recruited from the general population. Enrollment is restricted to the geographical area.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2023-04 (Actual); Study Completion 2023-04 (Actual)

PRIMARY OUTCOMES:
Follicle number per ovary | 1 day
  The number and size of all follicles in each ovary will be assessed by ultrasonography

SECONDARY OUTCOMES:
Follicle number per cross section | 1 day
  The number all follicles in a single cross sectional plane of each ovary will be assessed by ultrasonography
Ovarian volume | 1 day
  The size of each ovary will be determined by ultrasonography for each participant and compared across groups.
Stromal echogenicity on ultrasound | 1 day
  The brightness of the ovarian stroma in a single cross section will be determined by ultrasonography for each participant and compared across groups.
Ovarian area-stromal area ratio | 1 day
  The ratio of the stromal area to the total ovarian area of the ovary in a single cross section will be determined by ultrasonography for each participant and compared across groups.
LH-FSH ratio | 1 day
  The ratio of circulating LH to FSH concentrations in the serum will be determined for each participant and compared across groups
Hirsutism Score | 1 day
  Degree of hirsutism as judged by the Ferriman-Gallwey scale will be determined and compared across groups
Androgen concentrations | 1 day
  Total testosterone, androstenedione and free androgen index concentrations in serum will be determined and compared across groups.
Menstrual Cycle Length | 1 day
  Average menstrual cycle length as determined by self-reported history will be determined and compared across groups
Serum markers of metabolic syndrome | 1 day
  Lipids, glucose and HbA1C concentrations will be determined and compared across groups.
Blood Pressure | 1 day
  Blood pressure will be determined and compared across groups. [Time Frame: 1 day]
Body mass index | 1 day
  The ratio of weight to height will be determined and compared across groups.
Waist-to-hip ratio | 1 day
  The ratio of waist circumference to hip circumference will be determined and compared across groups
Body fat distribution | 1 day
  Percentage and distribution of fat and lean mass as assessed using DXA technology will be compared across groups.
Insulin sensitivity | 1 day
  Insulin sensitivity will be determined by administration of an oral glucose tolerance test and compared across groups.
Differences in diet composition assessed via food frequency questionnaire | 1 day
  A food frequency questionnaire will be administered to assess diet composition for the last three months and will be compared across groups
Differences in energy expenditure assessed via a waist-worn accelerometer | 1 week
  Participants will be asked to wear a small accelerometer device to assess physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Marla E Lujan, PhD, Principal Investigator — Cornell University; Steven Spandorfer, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Clinical and Translational Science Center, New York, New York, United States